CLINICAL TRIAL: NCT04728958
Title: Studying the Effect of Written Reflective Tasks With Healthcare Staff Working During the COVID-19 Health Pandemic
Brief Title: Reflective Tasks With Healthcare Workers During COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Collaborators: Sheffield Teaching Hospitals NHS Foundation Trust (Other); The Leeds Teaching Hospitals NHS Trust (Other); York Teaching Hospitals NHS Foundation Trust (Other); Bradford Teaching Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 170732
Record Dates: First submitted 2021-01-11; First posted 2021-01-28 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2021-01

CONDITIONS: Wellbeing; Psychological Distress; Emotional Distress; Depression; Happiness; Affect
Keywords: Gratitude
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: T-tests compare the mean differences between groups split across the two IVs (intervention & time), due to the between factors and within factors levels of the two IVs.
  Descriptive Statistics & t-tests will be used to compare and assess cumulative gratitude week-by-week
Who Masked: Participant
Masking Description: Participants will only be aware of the arm they are allocated to and not the other arms available. They will also be unaware as to whether this is a treatment arm or the comparator control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gratitude Journal (Experimental): Participants will be given instructions and asked to write a gratitude journal about their week, focusing upon what they are grateful for. Over the course of the 4-week intervention they will be asked to do this weekly (a total of four times).
  Interventions: Behavioral: Gratitude
- Weekly Diary (Placebo Comparator): Participants will be given instructions and asked to write a diary about their week, focusing upon both the good and the bad they have experienced that week. Over the course of the 4-week intervention they will be asked to do this weekly (a total of four times).
  Interventions: Behavioral: Gratitude

INTERVENTIONS:
Behavioral: Gratitude — A positive psychology intervention using expressions of gratitude
  Other Names: Gratitude Letter; Gratitude Diary; Gratitude Journal; Appreciation Letter; expressing gratitude; positive psychology intervention

SUMMARY:
The healthcare workforce is amongst the most stressed in the United Kingdom (UK). The Coronavirus (COVID-19) health pandemic has increased depression, anxiety, insomnia and distress in this population. Gratitude interventions have been shown to improve wellbeing, alongside reducing risk factors associated with the aforementioned mental health conditions. This online Randomised Control Trial of 219 healthcare staff, will investigate the effects of a gratitude intervention on wellbeing (gratitude, positive affect, happiness) and psychological distress (depression and negative affect). Means of pre- and post-outcome measures of two groups (gratitude journal and control) will be assessed for differences utilising t-tests.

DETAILED DESCRIPTION:
The healthcare workforce is amongst the most stressed in the UK, with 40.3% of staff feeling unwell as a result of work-related stress in the past year. This is steadily increasing each year, rising 3.5% from 36.8% since 2016. Chronic stress can cause psychological health problems, including low mood, anxiety and insomnia. Unfortunately, only 29.3% of staff across the NHS felt their trust took positive action on health and wellbeing, which may contribute to and prolong this continued rise in work-related stress.

With the COVID-19 health pandemic adding additional pressure to the NHS, healthcare workers (HCWs) are at further risk of mental health problems, including post-traumatic stress disorder, depression and substance misuse, as evident from historical health pandemics. Furthermore, preliminary data from China during the COVID-19 health pandemic indicated frontline HCWs experienced depression (50.4%), anxiety (44.6%), insomnia (34%) and distress (71.5%). A systematic review identified risk factors for increased psychological distress of HCWs during a health pandemic: being female, a nurse and experiencing stigmatised attitudes from the general public, as well as being quarantined. Perceived control and social support were associated with lower distress. Recommendations were made, to encourage a sense of autonomy (with information and resources), increase social support and to initiate public health campaigns with accurate facts, to reduce stigma and distress.

Positive Psychology Interventions (PPIs) are one approach for promoting autonomy and reducing distress, by increasing positive emotions, behaviours, and/or thoughts, thereby increasing the wellbeing of an individual. Positive psychology focuses on optimism, positive attitude and gratitude, to encourage creativity, improve happiness and reduce mental barriers to productivity, as opposed to focusing on 'problems'. PPIs include gratitude journals, using affirmations, strength focussing exercises and mindful meditations. PPIs in workplaces have improved performance, job wellbeing, engagement and other areas, whilst reducing negative performance and negative job wellbeing.

PPIs have focused on gratitude as a target for improving wellbeing, due to the inverse relationship found between gratitude and burnout. Burnout is a state of emotional and physical exhaustion, cynicism and detachment from work, caused by prolonged stress. Gratitude is a positive, social emotion, similar to appreciation, which can either be state (of being) or trait (dispositional). State gratitude is experienced when undeserved acts of kindness or generosity are given freely by another person. Whereas trait gratitude is viewed as a characteristic of a person, that varies in intensity and frequency throughout their daily life. Gratitude interventions have found improvements (with a small to medium effect size) in quality of relationships, wellbeing and optimism, alongside job satisfaction . Furthermore, a reduction in anxiety, depression and negative affect is also evident.

Gratitude interventions utilise both expression and self-reflection as their methodological properties. Expression includes giving small tokens of appreciation or paying gratitude visits. Self-reflection includes writing personal gratitude lists or journals. Gratitude lists were as effective as clinical therapies when working with excessive worry. Whereas, sharing a gratitude letter was not as effective at improving gratitude, furthermore expression of gratitude immediately induced feelings of embarrassment and discomfort. However, increases in elevation were noted here, namely improved job performance, connectedness, empowerment and autonomy. The reduced effectiveness of this expressive gratitude intervention, may be due to barriers in engagement with the intervention, including the expected awkwardness of the situation and the 'gratitude expresser's' mood.

Effectiveness of gratitude interventions in improving gratitude is likely to be affected by both traits of participants and specificities of the intervention, such as length. Research found trait gratitude moderated the effectiveness of the gratitude intervention in increasing gratitude. This supports the resistance hypothesis, suggesting that those who are predisposed to experience gratitude will not benefit from a gratitude intervention. Irrespective of gratitude moderation, wellbeing significantly improved. The duration of the intervention may also have an impact on effectiveness. Research found higher life satisfaction, more gratitude and an improved positive affect in HCWs, after writing a gratitude diary bi-weekly over 4-weeks. Whereas a shorter 5-day intervention in the workplace, using a similar journaling methodology, was not effective at improving gratitude. This may be explained by research, which found a cumulative improvement in gratitude and happiness over 8-weeks of grateful letter writing, indicating gratitude interventions are required to be of a reasonable length in order to be effective.

HCWs are suffering from psychological distress as a result of the COVID-19 health pandemic. It is vital interventions are offered to support their wellbeing. Gratitude interventions are effective at improving wellbeing and reducing psychological distress, namely the risk factors associated with psychological distress in HCWs at present. Self-reflective gratitude interventions, over a period of weeks are effective at improving gratitude with HCWs, without inducing embarrassment, discomfort or barriers to engagement. However, it is not clear if there are differences in effectiveness dependent upon the methodological properties of the intervention.

This study will aim to investigate the effects of a gratitude intervention with HCWs, with a view to increasing state gratitude and psychological wellbeing (subjective happiness and positive affect), whilst reducing psychological distress (negative affect and depression).

Objectives

1. To investigate if gratitude interventions are effective at increasing state gratitude in HCWs
2. To investigate if gratitude interventions are effective at reducing psychological distress and improving wellbeing in HCWs
3. To investigate if high baseline trait gratitude is a moderator of changes in state gratitude, psychological distress and wellbeing after a gratitude intervention

Hypotheses

1. A gratitude intervention will increase state gratitude in HCWs
2. A gratitude intervention will improve wellbeing (positive affect and subjective happiness) and reduce psychological distress (depression and negative affect) in HCWs
3. High levels of trait gratitude will moderate the outcomes

ELIGIBILITY:
Inclusion Criteria:

* Staff working in a healthcare environment during the COVID-19 health pandemic, in clinical or non-clinical roles
* Basic understanding of the English language

Exclusion Criteria:

* Those engaged in other research projects
* Those without access to an electronic device to complete measures on
* Those without access to an email address
* Those receiving any other form of psychological intervention
* People who cannot commit to engage in a 4-week intervention study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Change in Depression Level | Pre- to post-intervention (28 days)
  Patient Health Questionnaire-9 (PHQ-9). This 9-item questionnaire, uses a 4-point likert scale to measure depression level. Minimum score = 0; maximum score = 27. Higher scores indicate higher levels of depression. Positive change scores indicates a worse outcome.
Change in Subjective Happiness Level | Pre- to post-intervention (28 days)
  Subjective Happiness Scale (SHS). This 4-item questionnaire, uses a 7-point likert scale to measure happiness level. Minimum score = 7; maximum score = 28. Higher scores indicate higher subjective happiness levels. Positive change scores indicates a better outcome.

SECONDARY OUTCOMES:
Change in State Gratitude | Pre- to post-intervention (28 days)
  Gratitude Adjective Checklist (GAC). This 3-item measures of state gratitude uses a 5-point likert scale. Minimum score = 3; maximum score = 15. Higher scores indicate higher levels of state gratitude. A positive change score indicates a better outcome.
State Gratitude Score | Weekly (Day 1, Day 7, Day 14, Day 28)
  Gratitude Adjective Checklist (GAC). This 3-item measures of state gratitude uses a 5-point likert scale. Minimum score = 3; maximum score = 15. Higher scores indicate higher levels of state gratitude. A positive change score indicates a better outcome.
Change in Trait Gratitude | Pre- to post-intervention (28 days)
  The gratitude Questionnaire-6 (GQ-6). This 6-item measure of trait gratitude uses a 7-point likert scale. Minimum score = 6; maximum score = 42. Higher scores indicate higher levels of Trait gratitude. A positive change score indicates a better outcome.
Trait Gratitude score | Pre-intervention
  The gratitude Questionnaire-6 (GQ-6). This 6-item measure of trait gratitude uses a 7-point likert scale. Minimum score = 6; maximum score = 42. Higher scores indicate higher levels of Trait gratitude.

OTHER OUTCOMES:
Positive and Negative Affect | Weekly (Day 1, Day 7, Day 14, Day 28)
  The Positive and Negative Affect Scale - Short Form (PANAS-SF) is a 10-item measure of positive and negative affect. It uses a 5-point likert scale across both positive and negative affect. Positive affect is scored separately to negative affect, each with a minimum score of 5 and a maximum score of 25. High score on positive affect items indicate higher positive affect, whilst higher scores on negative affect items indicate higher negative affect.

CONTACTS AND LOCATIONS:
Overall Officials: Vicky Lamb, MSc, Principal Investigator — University of Sheffield
Locations (1):
- University of Sheffield, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD will be stored securely on the UniDrive, in a shared folder between the principal investigator and the research supervisor. Raw data will also be stored on the Qualtrics system, under a password protected log-in.
  Study results will be available in the University of Sheffield Online Research Data (ORDA) hub once completed. Sensitive and personal information will not be available as the key linking participant numbers to the personal will be destroyed once the study is completed. The data available will be completely anonymised.